CLINICAL TRIAL: NCT00490854
Title: A Crossover Study to Evaluate the Efficacy and Safety of Preprandial Human Insulin Inhalation Powder (HIIP) Compared to Once-Daily NPH in Insulin-Naïve Patients With Type 2 Diabetes Mellitus on Oral Agents
Brief Title: A Study for Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Alkermes, Inc. (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10513; H7U-JE-IDBF
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Last update posted 2008-07-10 (Estimated); Status verified 2008-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Human Insulin Inhalation Powder; Drug: Neutral protamine hagedorn insulin
- 2 (Experimental)
  Interventions: Drug: Human Insulin Inhalation Powder; Drug: Neutral protamine hagedorn insulin

INTERVENTIONS:
Drug: Human Insulin Inhalation Powder — patient specific, inhaled, at meals, 76 weeks
  Other Names: LY 041001
Drug: Neutral protamine hagedorn insulin — patient specific dose, injected, daily, 76 weeks

SUMMARY:
The purpose of the study is to compare the human insulin inhalation powder plus oral anti-hyperglycemic medication with injected insulin (neutral protamine hegedom insulin) plus oral anti-hyperglycemic medication on lowering the blood sugar level.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes mellitus for at least 6 months
2. One or more oral antihyperglycemic medications for at least 12 weeks
3. HbA1c equal to or greater than 7.0%, and equal to or less than 10.5%
4. Nonsmokers, have not smoked for at least 6 months and agree not to smoke (cigars, cigarettes, or pipes) or use smokeless tobacco for the duration of the study
5. Satisfactory lung function results to meet the requirement of the study

Exclusion Criteria:

1. Previously received any form of inhaled insulin
2. Have a current diagnosis or past history of asthma, chronic obstructive pulmonary disease or other clinically relevant lung disease
3. History or presence of liver disease
4. History or presence of kidney disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2007-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Mean change in Hemoglobin A1c (HbA1c) from baseline to the end of each treatment period of Primary Phase | 24, 48 and 76 weeks after Randomization

SECONDARY OUTCOMES:
8-point SMBG profiles. | 24, 48 and 76 weeks after Randomization
Mean change in HbA1c from baseline to the end. | 24, 48 and 76 weeks after Randomization
Mean dosage of both preprandial and basal insulin. | 24, 48 and 76 weeks after Randomization
Inhaler reliability. | 24, 48 and 76 weeks after Randomization
Patient-reported outcomes questionnaires. | 24, 48 and 76 weeks after Randomization

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- Japan (13):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukushima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gunma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shiga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toyama

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com